CLINICAL TRIAL: NCT02251236
Title: Elvitegravir (EVG) Cerebrospinal Fluid (CSF) Pharmacokinetics in HIV-Infected Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gilead Sciences (Industry); University at Buffalo (Other)
Responsible Party: Principal Investigator, Scott Letendre, Associate Professor of Medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-236-1266
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: Stribild; Genvoya; elvitegravir; Cerebrospinal Fluid; HIV
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Cobicistat; Emtricitabine; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stribild Arm (Other): Stribild Arm is for participants taking Stribild at the time of study entry. Participants taking Stribild at the time of study entry will switch to Genvoya before the second PK.
  Interventions: Drug: Stribild; Drug: Genvoya
- Genvoya Arm (Other): Genvoya Arm is for participants already taking Genvoya at the time of study entry. Participants taking Genvoya at the time of study entry will continue Genvoya for the second PK.
  Interventions: Drug: Genvoya
- Untreated Arm (Other): Untreated Arm is for participants who are not taking ART at the time of study entry. Participants will start Stribild at entry and switch to Genvoya before the second PK.
  Interventions: Drug: Stribild; Drug: Genvoya

INTERVENTIONS:
Drug: Stribild — To be administered orally, once daily with food.
  Other Names: Co-formulated elvitegravir/ cobicistat/ emtricitabine/ tenofovir disoproxil fumarate
  Arms: Stribild Arm; Untreated Arm
Drug: Genvoya — To be administered orally, once daily with food.
  Other Names: Co-formulated elvitegravir/ cobicistat/ emtricitabine/ tenofovir alafenamide

SUMMARY:
The project will have two tracks, one for participants who are currently taking elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate or E/C/F/tenofovir alafenamide (E/C/F/TDF or E/C/F/TAF) single-tablet regimen* (STR) (Track A) and one for participants who will begin therapy with E/C/F/TDF or E/C/F/TAF STR during the study (Track B).

Participants will take E/C/F/TDF and/or E/C/F/tenofovir alafenamide fumarate (E/C/F/TAF) STR** (if available) for 24 weeks.

*Co-formulation of 150 mg of elvitegravir, 150 mg of cobicistat, 200 mg of emtricitabine, and 300 mg of tenofovir disoproxil fumarate.

**Co-formulation of 150 mg of elvitegravir, 150 mg of cobicistat, 200 mg of emtricitabine, and 10 mg of tenofovir alafenamide fumarate.

DETAILED DESCRIPTION:
The proposed project will be a prospective, open-label treatment trial of 14 HIV-infected adults. Participants will be enrolled in two tracks. Track A will enroll participants who have been taking E/C/F/TDF to E/C/F/TAF for at least 12 weeks. Track B will enroll participants who are not taking ART and no prior exposure to elvitegravir and no genotypic drug resistance to any component of E/C/F/TDF to E/C/F/TAF. CSF and blood will be collected twice in Track A (two on-treatment assessments) and three times in Track B (one pre-treatment, two on-treatment assessments). If possible, we plan to time assessments to bridge the transition from E/C/F/TDF to E/C/F/TAF so that all participants will ideally have one CSF collection on each regimen, enabling a paired comparison of tenofovir concentrations between the two tenofovir formulations. We estimate that 28 on-treatment CSF collections will be sufficient to provide a small-sample estimate of the distribution of elvitegravir, tenofovir and TAF into CSF.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18-60 years. Able and willing to provide informed consent.
* Presence of HIV-1 infection as documented by a licensed ELISA test kit and confirmed by Western blot or HIV RNA.
* Track A (Currently taking E/C/F/TDF or E/C/F/TAF): Taking E/C/F/TDF or E/C/F/TAF for at least 3 months prior to screening and undetectable plasma HIV-1 RNA (≤ 40 copies/mL)
* Track B (Currently not taking ART): Off ART for at least 3 months. Prior exposure to TDF and FTC will be allowed but subjects must not have primary genotypic drug resistance mutations to elvitegravir, tenofovir, or emtricitabine (see Exclusion Criteria)
* Plasma HIV-1 RNA ≥ 5,000c/mL and CD4+ T-cell count ≥200cells/mm3.

Exclusion Criteria:

* Track B: Presence of primary drug resistance mutations for EVG, tenofovir, or emtricitabine.
* Use of drugs of abuse or alcohol which would interfere with adherence or completion of this study. While on-study, subjects will be instructed not to consume alcohol for 48 hours prior to pharmacokinetic sampling days.
* Pregnancy or breast-feeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to study entry and day of entry.
* Chronic, severe, or other medical conditions that, in the opinion of the investigator, would interfere with the subjects ability to participate in the protocol.
* Use of prohibited protocol-specified drugs, prescription or over-the-counter, within 14 days prior to study entry.
* Bleeding abnormality or other contraindication to lumbar puncture.
* Moderate or severe cognitive impairment by history or based on Montreal Cognitive Assessment.
* Hepatitis B surface antigen (HBsAg) positive (Positive anti-HBs antibody and negative HBsAg results are acceptable)
* Hepatitis C antibody (HCV Ab) positive
* Laboratory parameters documented within 21 days prior to study entry that would increase the risk for adverse events:

  1. Hemoglobin < 12.5 g/dL for men; < 11.5 g/dL for women;
  2. Platelet count < 100,000 platelets/mm3;
  3. AST (SGOT) or ALT (SGPT) > 1.5 x the upper limit of normal (ULN);
  4. Estimated GFR<70 ml/min
  5. Weight less than 50 kg

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Letendre, MD, Principal Investigator — UCSD
Locations (1):
- UC San Diego AntiViral Research Center, San Diego, California, United States

REFERENCES:
- [Derived] Ma Q, Ocque AJ, Morse GD, Sanders C, Burgi A, Little SJ, Letendre SL. Switching to Tenofovir Alafenamide in Elvitegravir-Based Regimens: Pharmacokinetics and Antiviral Activity in Cerebrospinal Fluid. Clin Infect Dis. 2020 Aug 14;71(4):982-988. doi: 10.1093/cid/ciz926. PMID 31560741

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
Started | 9 | 5 | 0
Completed | 9 | 5 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants enrolled in the Untreated Arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm | Total
Number analyzed (Participants) | 9 | 5 | 0 | 14
Age, Continuous [Median (Full Range); unit: years] | 34 [23 to 56] | 45 [32 to 50] |  | 34.5 [23 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  | 1
  Male | 8 | 5 |  | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 1 |  | 2
  White | 8 | 4 |  | 12
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Plasma HIV RNA ≤ 40 copies/mL [Count of Participants; unit: Participants] | 9 | 5 |  | 14
CD4+ T-cell Count [Median (Full Range); unit: cells/µL] | 601 [502 to 1071] | 784 [262 to 944] |  | 717 [262 to 1071]

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Elvitegravir in Cerebrospinal Fluid at Baseline
Time Frame: Baseline
Population: No participants enrolled in the Untreated Arm
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
Number analyzed (Participants) | 9 | 5 | 0
ng/mL | 4.3 [3.11 to 5.20] | 2.72 [1.75 to 3.48] |

2. Primary Outcome: Concentration of Elvitegravir in Cerebrospinal Fluid at Week 24
Time Frame: Week 24
Population: No participants enrolled in the Untreated Arm
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
Number analyzed (Participants) | 9 | 5 | 0
ng/mL | 5.90 [4.44 to 6.60] | 3.09 [3.02 to 3.62] |

3. Primary Outcome: Concentration of Tenofovir in Cerebrospinal Fluid at Baseline
Time Frame: Baseline
Population: No participants enrolled in the Untreated Arm
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
Number analyzed (Participants) | 9 | 5 | 0
ng/mL | 3.03 [2.13 to 4.84] | 0.49 [0.35 to 0.67] |

4. Primary Outcome: Concentration of Tenofovir in Cerebrospinal Fluid at Week 24
Time Frame: Week 24
Population: No participants enrolled in the Untreated Arm
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
Number analyzed (Participants) | 9 | 5 | 0
ng/mL | 0.507 [0.344 to 1.197] | 0.481 [0.255 to 0.556] |

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: No participants enrolled in the Untreated Arm so the number of participants at risk is zero
Arm/Group | Stribild Arm | Genvoya Arm | Untreated Arm
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 4/9 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stribild Arm (N=9) | Genvoya Arm (N=5) | Untreated Arm (N=0)
Headache, Grade 3 (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine Clearance Reduction, Grade 3 (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stribild Arm (N=9) | Genvoya Arm (N=5) | Untreated Arm (N=0)
Elevated Hepatic Alanine Transaminase, Grade 1 (Hepatobiliary disorders) | 1 (2) | 1 (1) | 0 (0)
Elevated Serum Glucose, Grade 1 (Endocrine disorders) | 1 (2) | 1 (1) | 0 (0)
Elevated Lactic Acid, Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia, Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated Serum Bicarbonate, Grade 1 (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Elevated Creatine Kinase, Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated Serum Creatinine, Grade 1 or 2 (Renal and urinary disorders) | 1 (3) | 1 (1) | 0 (0)
Hypernatremia, Grade 2 (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Hepatic Aspartate Transaminase, Grade 2 (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT02251236/Prot_SAP_000.pdf